CLINICAL TRIAL: NCT00784849
Title: Pilot Trial to Determine the Feasibility of a One Step Sentinel Lymph Node Biopsy Procedure Using Radiolabeled Methylene Blue (IND 70,627)
Brief Title: Feasibility of One-Step Sentinel Lymph Node (SLN) Biopsy With Radiolabeled Methylene Blue (IND 70,627)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, Varney Rannells, Research Coordinator, Louisiana State University Health Sciences Center in New Orleans
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LSU #6169
Record Dates: First submitted 2008-11-03; First posted 2008-11-04 (Estimated); Results first posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; diagnostic; lymph nodes
MeSH Terms: conditions — Breast Neoplasms; Disease | interventions — Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): One arm diagnostic
  Interventions: Drug: Methylene blue

INTERVENTIONS:
Drug: Methylene blue — 1 mC1
  Other Names: SNL biopsy; breast cancer biopsy

SUMMARY:
The purpose of this study is to develope a one-step procedure to perform a biopsy of axillary lymph nodes on the same side as the breast tumor in women diagnosed with breast cancer.

DETAILED DESCRIPTION:
This study proposes the use of a newly developed experimental radioactive dye (radiolabeled methylene blue). On the day of surgery, the patient receives a single injection of the experimental radioactive dye after anesthesia. The injection will be in the location around the breast tumor. The surgeon makes a small cut in the armpit on the side of the cancer and is able to locate the lymh nodes that collect drainage from the cancerous area by detecting lymph nodes with higher radioactivity using a hand-held detector (a Geiger counter-like device) and/or visually identifying lymph nodes stained blue by the dye. These lymph nodes are then removed and analyzed by pathologists for the presence of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Stage 0,I, II breast cancer
* Clinical node status N0, N1
* No know allergy to iodine, lymphazurin or methylene blue dyes

Exclusion Criteria:

* Patient cannot be pregnant or nursing
* Prisoners will not be eligible
* Women under the age of 18 will not be eligible
* Patients with a known allergy to iodine or methylene blue or lymphazurin blue dyes

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene A Woltering, MD, Principal Investigator — LSU Health Sciences Center - New Orleans LA
Locations (2):
- United States (2):
  - University Medical Center, Lafayette, Louisiana
  - LSU Interim Hospital, New Orleans, Louisiana

RESULTS

PARTICIPANT FLOW:
Groups:
- Sentinel Lymph Node Biopsy With Radiolabeled Methylene Blue: One arm diagnostic using 1 mCi of 125-I Methylene blue dye to find sentinel lymph nodes
Period: Overall Study
Arm/Group | Sentinel Lymph Node Biopsy With Radiolabeled Methylene Blue
Started | 62
Completed | 62
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sentinel Lymph Node Biopsy With Radiolabeled Methylene Blue
Number analyzed (Participants) | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 62

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants That Have Sentinel Nodes Which Are Radioactive or Blue, or Radioactive and Blue or Have Efferent Blue Lymphatics Leading up to the Sentinel Node(s)
Time Frame: intraoperatively; up to 6 hours
Measure: Number; unit: participants
Arm/Group | Sentinel Lymph Node Biopsy With Radiolabeled Methylene Blue
Number analyzed (Participants) | 62
participants
  Radioactive | 58
  Blue | 55
  Radioactive and Blue | 55
  Efferent blue lymphatics leading up to the SLN | 0

2. Secondary Outcome: Safety (Allergic Reaction to Blue Dye)
Description: number of participants who had a systemic allergic reaction such as hives, shortness of breath, hypotension
Time Frame: intraoperatively up to 6 hours
Measure: Number; unit: participants
Arm/Group | Sentinel Lymph Node Biopsy With Radiolabeled Methylene Blue
Number analyzed (Participants) | 62
participants | 0

3. Secondary Outcome: Superficial Skin Necrosis
Description: the number of participants who developed post-operative skin necrosis within 2 weeks of surgery
Time Frame: 2 weeks postoperatively
Measure: Number; unit: participants
Arm/Group | Sentinel Lymph Node Biopsy With Radiolabeled Methylene Blue
Number analyzed (Participants) | 62
participants | 2

ADVERSE EVENTS:
Arm/Group | Sentinel Lymph Node Biopsy With Radiolabeled Methylene Blue
Serious Adverse Events (participants affected / at risk) | 0/62
Other Adverse Events (participants affected / at risk) | 2/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sentinel Lymph Node Biopsy With Radiolabeled Methylene Blue (N=62)
superficial skin necrosis (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes